CLINICAL TRIAL: NCT06509997
Title: MRG003 Combined With Dalpicicilip Posterior Line in the Treatment of Recurrent/Metastatic CDKN2A Gene Variant Head and Neck Squamous Cell Carcinoma: A Phase II Clinical Trial
Brief Title: A Phase II Study of Anti-EGFR Antibody-drug Conjugate (ADC) Combine With CDK4/6 Inhibitors Posterior Line in the Treatment of Recurrent/Metastatic CDKN2A Gene Variant Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Liu (Other)
Responsible Party: Sponsor-Investigator, Lei Liu, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-HNC-II-006
Record Dates: First submitted 2024-07-10; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Recurrent/metastatic head and neck squamous cell carcinoma; CDKN2A gene variant; CDK4/6 inhibitor; Antibody-drug conjugate; EGFR inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: A single-arm Phase II clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG003+Dalpicicilip (Experimental): Patients meeting the inclusion criteria were given MRG003 (D1, IVGTT, Q3W) in combination with Darcilil (D1-21, PO, Q4W) after completing the relevant pre-treatment examination until progression or intolerable toxicity occurred.
  Interventions: Drug: MRG003 combined with Dalpicicilip

INTERVENTIONS:
Drug: MRG003 combined with Dalpicicilip — MRG003, intravenous infusion, D1, once every 3 weeks; Dalpicicilip, taking orally, D1-21, once every 4 weeks, maintain use until progression or emergence of intolerable toxicity.

SUMMARY:
A Single-arm, Phase II Study of MRG003 combined with Dalpicicilip posterior line in the treatment of recurrent/metastatic CDKN2A gene variant head and neck squamous cell carcinoman (HNSCC). The objective of this study was to evaluate the safety and efficacy of MRG003 combined with the Dalpicicilip posterior line in the treatment of recurrent/metastatic CDKN2A gene variant HNSCC.

DETAILED DESCRIPTION:
In this study, patients meeting the inclusion criteria were given MRG003 (D1, IVGTT, Q3W) in combination with Darcilil (D1-21, PO, Q4W) after completing the relevant pre-treatment examination until progression or intolerable toxicity occurred. Objective response rate and safety will be the primary outcome measures. Adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤75 years old;
2. Patients with recurrent or metastatic head and neck squamous cell carcinoma (including oral cavity, oropharynx, hypopharynx, larynx, etc.) confirmed by histology or cytology, recurrent patients cannot receive local treatment such as surgery or radiotherapy, and have failed to receive PD-1 (L1) inhibitors and/or platinum drugs in the past, which can be first-line combination regimens or sequential administration. Progression after receiving PD-1 (L1) inhibitors and/or platinum-based drugs;
3. Receive ≤2 lines of treatment;
4. ECOG score 0~1;
5. Lack of CDKN2A function;
6. At least one evaluable lesion according to RECIST (version 1.1) criteria;
7. Adequate organ function;
8. The expected survival time is greater than 3 months;
9. No serious organic heart disease or arrhythmia;
10. Women of childbearing age (15-49 years) must undergo a pregnancy study within 7 days before starting treatment and the results are negative; Fertile men and women must consent to the use of effective contraception to ensure that they do not become pregnant during the study period and for 3 months after stopping treatment;
11. Obtain the "informed consent" voluntarily signed by the patient.

Exclusion Criteria:

1. ≥ grade 2 peripheral neuropathy (according to CTCAE 5.0).
2. Surgery or any other form of systemic or local anti-tumor therapy, including maintenance therapy or radiotherapy for head and neck squamous cell carcinoma (including palliative care, except palliative care for non-target lesions), is expected to be required during the study period.
3. Systematic chemotherapy was received within 3 weeks before the first administration of the drug, small molecule targeted therapy was received within 2 weeks before the first administration or 5 half-lives (depending on the time), antitumor biotherapy, macromolecule targeted therapy or immunotherapy was received within 4 weeks before the first administration of the drug. Or major surgery (except minor surgery performed within 2 weeks and complete recovery); Radiotherapy was received within 14 days prior to initial administration of the investigational drug (except for central nervous system radiotherapy, which required a washout period of ≥28 days).
4. Known to have active central nervous system metastasis and/or cancerous meningitis. Patients with treated BMS may participate in the study if their condition is stable and they do not:

   * Progressive or new neurological deficits, seizures, evidence of increased intracranial pressure, vomiting, or headache;
   * MRI shows evidence of enlargement at least 4 weeks before first dosing and at least 14 days before study drug dosing Corticosteroids are required.
5. Residual toxic effects (except alopecia, fatigue and grade 2 hypothyroidism) caused by previous antitumor therapy (including immunotherapy, targeted therapy, chemotherapy or radiotherapy) or clinically significant laboratory test outliers higher than grade 1 (CTCAE v5.0).
6. Uncontrolled or poorly controlled heart disease, including a history of congestive heart failure (CHF) ≥2 (CTCAE v5.0 or New York Heart Association rating), myocardial infarction, unstable angina, ventricular tachycardia or tip twisting ventricular tachycardia, or arrhythmias requiring treatment within the 6 months prior to admission, For example, men with QTcF > 450 ms and women with QTcF > 470 ms have complete left bundle branch block or third-degree atrioventricular block. QTcF= QT/ (RR^0.33).
7. Pulmonary embolism or deep vein thrombosis (except for catheter-derived thrombosis at infusion port or PICC) occurred within 3 months prior to the first administration of the drug.
8. There is a known prior history of malignancy (except in patients with basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, carcinoma in situ, or papillary carcinoma of the thyroid who have undergone radical surgery), unless the patient has received potentially curable therapy and has been free of disease recurrence for 5 years since starting treatment. Note: The 5-year recurrence-free time requirement does not apply to head and neck squamous cell carcinoma in patients enrolled in this trial.
9. Any serious or uncontrolled systemic disease, including uncontrolled or poorly controlled hypertension (such as systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg), glycosuria (glycated blood red and egg white (HbA1c) >8%), etc.
10. Patients with a history of active bleeding, clotting disorders, or receiving coumarin anticoagulant therapy.
11. Known allergic reactions to any component or excipient of MRG003 (citric acid monohydrate, sodium citrate dihydrate, trehalose dihydrate, sodium chloride and polysorbate 80), or grade ≥3 allergic reactions to other prior anti-EGFR drugs (including investigational drugs) or to other monoclonal antibodies.
12. Known active hepatitis B or C. Active hepatitis B is defined as known HBsAg positive and HBV DNA≥500 IU/mL. Active hepatitis C is defined as a known positive hepatitis C antibody and a known quantitative hepatitis C virus HCV RNA result greater than the lower limit of detection. Other serious liver diseases are present, including chronic autoimmune liver disease, primary biliary cirrhosis or sclerosing cholangitis, alcoholic liver disease, or non-alcoholic steatohepatitis (NASH).
13. Concurrent severe, uncontrolled infection or known human immunodeficiency virus (HIV) (HIV antibody positive) infection, or a diagnosis of acquired immune deficiency syndrome (AIDS); Or uncontrolled autoimmune disease; Have previously received an allogeneic tissue/organ transplant, stem cell or bone marrow transplant, or have previously received a solid organ transplant.
14. Active bacterial, viral, fungal, rickettsial, or parasitic infections requiring systemic anti-infective therapy (unless treatment is obtained and resolves prior to administration of the investigational drug).
15. The live virus vaccine was administered within 30 days prior to the first administration of the investigational drug. Seasonal influenza vaccines or approved COVID-19 vaccines that allow the use of inactivated viruses must be at least one week from the time of first administration.
16. A history of interstitial pneumonia, severe chronic obstructive pulmonary disease with respiratory failure, severe pulmonary insufficiency, and symptomatic bronchospasm.
17. Immunological based treatment for any reason, including long-term use of a systemic steroid equivalent to >10 mg/ day of prednisone within 7 days before the first administration of the study drug or at any time during study participation. Note: Inhaled or topical steroids or systemic corticosteroids equivalent to ≤10 mg/ day of prednisone are permitted, as are short-term corticosteroids equivalent to >10 mg/ day of prednisone (e.g., prodromal administration before contrast agent administration).
18. Uncontrolled pleural, abdominal, pelvic or pericardial effusions require drainage ≥ once a month.
19. Patients who have tested positive for pregnancy or are breastfeeding. Women and men who do not plan to use adequate contraception during treatment and within 180 days after the last treatment.
20. Any other illness or clinically significant laboratory parameter abnormality, serious medical or psychiatric illness/condition, and substance abuse, including alcohol abuse, that the investigator believes could compromise patient safety, study integrity, affect patient participation in the study or interfere with the purpose of the study and analysis of the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | approximately 9-10 weeks after start of study treatment
  Objective response rate
Safety and Tolerability | approximately 9-10 weeks after start of study treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
OS | 2 years
  overall survival
PFS | 1-2years
  Progression Free Survival
DOR | 1-2years
  Duration of response
DCR | 2 years
  Disease control rates